CLINICAL TRIAL: NCT01026142
Title: A Multicenter Randomized Phase III Study to Compare the Combination Trastuzumab and Capecitabine, With or Without Pertuzumab, in Patients With HER2-Positive Metastatic Breast Cancer That Have Progressed After One Line of Trastuzumab-Based Therapy in the Metastatic Setting (PHEREXA)
Brief Title: A Study of a Combination of Trastuzumab and Capecitabine With or Without Pertuzumab in Patients With HER2-positive Metastatic Breast Cancer (PHEREXA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MO22324; 2008-006801-17 (EudraCT Number)
Record Dates: First submitted 2009-11-27; First posted 2009-12-04 (Estimated); Results first posted 2016-10-13 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; pertuzumab; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A: Capecitabine + Trastuzumab (Active Comparator)
  Interventions: Drug: Capecitabine; Drug: Trastuzumab
- B: Capecitabine + Trastuzumab + Pertuzumab (Experimental)
  Interventions: Drug: Capecitabine; Drug: Pertuzumab; Drug: Trastuzumab

INTERVENTIONS:
Drug: Capecitabine — 1000 mg/m2 po twice daily for 14 days every 3 weeks
  Other Names: Xeloda
  Arms: B: Capecitabine + Trastuzumab + Pertuzumab
Drug: Capecitabine — 1250 mg/m2 po twice daily for 14 days every 3 weeks
  Other Names: Xeloda
  Arms: A: Capecitabine + Trastuzumab
Drug: Pertuzumab — 840 mg iv loading, then 420 mg iv every 3 weeks
  Other Names: Perjeta
  Arms: B: Capecitabine + Trastuzumab + Pertuzumab
Drug: Trastuzumab — 8 mg/kg iv loading, then 6 mg/kg iv every 3 weeks
  Other Names: Herceptin

SUMMARY:
This randomized, two-arm study evaluated the efficacy and safety of a combination of trastuzumab and capecitabine with or without pertuzumab in patients with human epidermal growth factor receptor 2 (HER2)-positive metastatic breast cancer. The study population consisted of female patients, whose disease had progressed during or following previous trastuzumab therapy for metastatic disease. All patients in Arm A and Arm B received trastuzumab (8 mg/kg iv as loading dose and then 6 mg/kg iv every 3 weeks thereafter) and capecitabine oral twice daily for 14 days every 3 weeks (1250 mg/m2 twice daily in Arm A and 1000 mg/m2 twice daily in Arm B). In addition, patients in Arm B received pertuzumab (840 mg iv as loading dose and then 420 mg iv thereafter) every 3 weeks. Study treatment continued until disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patients >/=18 years of age
* Metastatic HER2 positive breast cancer
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Disease progression during or following trastuzumab-based therapy for 1st line metastatic breast cancer (trastuzumab must have been part of the last prior treatment regimen)
* Prior treatment with taxane-containing regimen
* Left ventricular ejection fraction (LVEF) >/=50 percent
* For women of childbearing potential agreement to use highly effective non-hormonal form of contraception or two effective forms of non-hormonal contraception by patient and/or partner. Contraception must continue for duration of study treatment and for at least 6 months after last dose of study drug treatment

Exclusion Criteria:

* Prior treatment with pertuzumab or capecitabine
* Concurrent treatment with other experimental drug
* Concurrent immunotherapy or anticancer hormonal therapy
* Serious concurrent disease (e.g. active infection, uncontrolled hypertension, cardiovascular disease)
* Central nervous system (CNS) metastases, which are not well controlled
* History of exposure to anthracycline cumulative dose equivalent to 360mg/m2
* History of congestive heart failure of any New York Heart Association criteria, or serious cardiac arrhythmia requiring treatment
* History of myocardial infarction within 6 months prior to randomization
* History of LVEF decline to below 50% during or after prior trastuzumab therapy or other cardiac toxicity during previous trastuzumab treatment that necessitated discontinuation of trastuzumab
* History of another cancer which could affect compliance or result interpretation
* Inadequate organ function
* Pregnant or breastfeeding women
* life expectancy < 12 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2010-01-26 (Actual); Primary Completion 2015-05-29 (Actual); Study Completion 2017-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (190):
- Argentina (6):
  - Fundación Investigar, Buenos Aires
  - Hospital Britanico; Oncologia, Buenos Aires
  - Instituto FIDES, La Plata
  - Instituto de Investigaciones Clínicas Quilmes, Quilmes
  - Instituto de Oncología de Rosario, Rosario
  - ISIS Clinica Especializada, Santa Fe
- Austria (4):
  - A.Ö. Landesschwerpunktkrankenhaus Krems; Abtl. F. Innere Med., Krems
  - Landeskrankenhaus Rankweil; Interne E, Rankweil
  - Lkh Salzburg - Univ. Klinikum Salzburg; Iii. Medizinische Abt., Salzburg
  - Medizinische Universität Wien; Univ.Klinik für Innere Medizin I - Abt. für Onkologie, Vienna
- Belgium (11):
  - Imeldaziekenhuis, Bonheiden
  - AZ KLINA, Brasschaat
  - UZ Brussel, Brussels
  - GHdC Site Notre Dame, Charleroi
  - CH Jolimont - Lobbes (Jolimont), Haine-Saint-Paul
  - Jessa Zkh (Campus Virga Jesse), Hasselt
  - AZ Groeninge, Kortrijk
  - CHU Sart-Tilman, Liège
  - Clinique Saint-Joseph, Liège
  - Clinique Ste-Elisabeth, Namur
  - AZ Nikolaas (Lodewijk), Sint-Niklaas
- Brazil (5):
  - Oncologia Sul Capixaba Servicos Medicos - Oncosul, Cachoeiro de Itapemirim, Espírito Santo
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital Perola Byington, São Paulo, São Paulo
  - Hospital A. C. Camargo; Oncologia, São Paulo, São Paulo
  - Centro Oncológico de Mogi das Cruzes, São Paulo- SP, São Paulo
- Canada (3):
  - Durham Regional Cancer Centre, Oshawa, Ontario
  - Humber River Hospital, Toronto, Ontario
  - University Health Network; Princess Margaret Hospital; Medical Oncology Dept, Toronto, Ontario
- Uni Hospital For Tumours; Dept of Medical Oncology, Zagreb, Croatia
- Czechia (4):
  - Masarykuv onkologicky ustav; Oncology II, Brno
  - University Hospital; Oncology and Radiotherapy, Hradec Králové
  - Fakultni Poliklinika Vseobecne Fakultni Niemocnice; Onkologicka Klinika, Prague
  - Lekarske Fakulty Univerzity Karlovy Fakultni Nemocnice Na Bulovce; Ustav Radiacni Onkologie, Prague
- Estonia (2):
  - North Estonia Medical Centre Foundation; Oncology Centre, Tallinn
  - Tartu University Hospital; Clinic of Hematology and Oncology, Tartu
- France (15):
  - C.H. Du Pays D'aix En Provence Service du Dr Blanc, Aix-en-Provence
  - Centre Oncologie Du Pays Basque, Bayonne
  - Centre Hospitalier Fleyriat; Oncologie/Hematologie, Bourg-en-Bresse
  - CHU Henri Mondor; Service d'Oncologie Medicale, Créteil
  - Centre Georges Francois Leclerc; Oncologie 3, Dijon
  - Centre Leon Berard; Oncologie Genetique, Lyon
  - Centre Antoine Lacassagne; Hopital De Jour A2, Nice
  - Institut Curie; Oncologie Medicale, Paris
  - Hopital Saint Antoine; Sce Oncologie, Paris
  - Institut Jean Godinot; Oncologie Medicale, Reims
  - Centre Henri Becquerel; Oncologie Medicale, Rouen
  - Centre Rene Huguenin; CONSULT SPECIALISEES, Saint-Cloud
  - Hopital Hautepierre; Hematologie Oncologie, Strasbourg
  - Institut Claudius Regaud; Departement Oncologie Medicale, Toulouse
  - Clinique Pasteur; Oncologie Medicale, Toulouse
- Germany (25):
  - CAMPUS CHARITÉ MITTE; Tagesklinik für Onkologie u.Hämatologie, Berlin
  - Klinikum Sindelfinden Boblingen, Böblingen
  - Klinikum Bremen-Mitte gGmbH; Frauenklinik, Bremen
  - St. Elisabeth Krankenhaus Köln GmbH; Gynäkologie und Geburtshilfe, Cologne
  - Klinikum Darmstadt GmbH; Med. Klinik V; Onkologie & Hämatologie, Darmstadt
  - Klinikum Dortmund gGmbH Klinikzentrum Mitte, Dortmund
  - Universitätsklinikum Essen; Zentrum Für Frauenheilkunde, Essen
  - Klinikum Frankfurt Höchst GmbH; Klinik für Gynäkologie und Geburtshilfe, Frankfurt
  - Klinik Fulda, Medizinisches Versorgungszentrum Osthessen GmbH, Fulda
  - Universitätsklinikum Hamburg-Eppendorf; Zentrum für operative Medizin Klinik für Gynäkologie, Hamburg
  - HOPA MVZ GmbH, Hamburg
  - Diakovere Henriettenstift, Frauenklinik, Hanover
  - Medizinische Hochschule Zentrum Frauenheilkunde Abt.Gynäkologische Onkologie, Hanover
  - ViDia Christliche Kliniken Karlsruhe, Vincentius-Diakonissen-Kliniken gAG; Frauenklinik, Karlsruhe
  - Systemedic Frauenarzte Pruener Gang, Kiel
  - Institut für Versorgungsforschung in der Onkologie GbR Koblenz, Koblenz
  - Universitätsklinikum Schleswig-Holstein / Campus Lübeck; Klinik für Frauenheilkunde und Geburtshilfe, Lübeck
  - St. Vincenz-Elisabeth-Hospital; Katholisches Klinikum Mainz, Mainz
  - Klinikum rechts der Isar der TU München; Frauenklinik & Poliklinik, München
  - Universitätsklinikum Münster; Klinik für Frauenheilkunde und Geburtshilfe, Münster
  - St. Josefs Klinik; Medizinische Klinik, Offenburg
  - Praxis für Onkologie und Hämatologie, Recklinghausen
  - Johanniter Klinik, Stendal
  - Klinikum Mutterhaus der Borromaeerinnen gGmbH; Haematologie/Onkologie, Trier
  - GRN Klinik Weinheim, Weinheim
- Hong Kong (3):
  - Queen Mary Hospital; Surgery, Hong Kong
  - Queen Elizabeth Hospital; Clinical Oncology, Hong Kong
  - Tuen Mun Hospital; Clinical Oncology, Hong Kong
- Hungary (15):
  - Ogyi, Orszagos Gyogyszereszeti Intezet, Budapest
  - Semmelweis Egyetem Onkologiai Központ, Budapest
  - Fövárosi Önkormányzat Bajcsy-Zsilinszky Kórház; Onkológiai Osztály, Budapest
  - Orszagos Onkologiai Intezet; B Belgyogyaszati Osztaly, Budapest
  - Semmelweis Egyetem Aok; Iii.Sz. Belgyogyaszati Klinika, Budapest
  - Municipal Hospital of Uzsoki Utca; Centre of Oncoradiology, Budapest
  - Hospital of Aladar Petz; Dept of Oncoradiology, Győr
  - Békés Megyei Pándy Kálmán Kórház; Onkologiai tanszek, Gyula
  - Kaposi Mor County Hospital; Dept. of Oncology, Kaposvár
  - Borsod-Abauj-Zemplen Megyei Korhaz Es Egyetemi Oktato Korhaz; Onkologiai Osztaly, Miskolc
  - Josa Andras Korhaz; Dept of Oncoradiology, Nyíregyháza
  - Pécsi Tudományegyetem Áok; Onkoterapias Intezet, Pécs
  - Szegedi Tudomanyegyetem, AOK, Szent-Gyorgyi Albert Klinikai Kozpont, Onkoterapias Klinika, Szeged
  - Fejér Megyei Szent György Kórház; Onkológiai Osztály, Székesfehérvár
  - Jász-Nagykun-Szolnok Megyei Hetényi Géza Kórház; Onkológiai Osztály, Szolnok
- Italy (21):
  - Istituto Tumori Fondazione Pascale; Endocrinologia Oncologica, Napoli, Campania
  - Az. Osp. S. Orsola Malpighi; Istituto Di Oncologia Seragnoli, Bologna, Emilia-Romagna
  - Ospedale Cervesi di Cattolica ; Unità Operativa di Oncologia ed Oncoematologia, Cattalica, Emilia-Romagna
  - AUSL Cesena; Servizio di Oncologia, Cesena, Emilia-Romagna
  - Ausl Ravenna-Osp.Infermi; Day Hospital Oncologia Medica, Faenza, Emilia-Romagna
  - Ospedale Umberto I ASL di Ravenna Presidio Ospedaliero di Lugo, Lugo, Emilia-Romagna
  - Azienda USL di Ravenna; Unità Operativa di Oncologia Medica, Ravenna, Emilia-Romagna
  - Ospedale Infermi Di Rimini; Unità Operativa di Oncologia e Oncoematologia, Rimini, Emilia-Romagna
  - Istituto Regina Elena; Oncologia Medica A, Rome, Lazio
  - Uni Cattolica Policlinico Gemelli; Oncologia Medica Ist. Medicina Interna, Rome, Lazio
  - Asst Papa Giovanni XXIII; Oncologia Medica, Bergamo, Lombardy
  - ASST DI CREMONA; Dipartimento Aziendale Oncologico, Cremona, Lombardy
  - Ospedale Mater Salutis; Dept of Oncology, Legnago, Lombardy
  - ASST DI MONZA; Oncologia Medica, Monza, Lombardy
  - IRCCS Fondazione Maugeri; Oncologia Medica II, Pavia, Lombardy
  - ASST LARIANA; Oncologia, S. Fermo Della Battaglia (CO), Lombardy
  - A.O. Città della Salute e della Scienza - Presidio Molinette; divisione oncologia medica, Turin, Piedmont
  - Ospedale Civile; Oncologia Medica, Sassari, Sardinia
  - ARNAS-Ospedale Civico Maurizio Ascoli; Unità Operativa di Oncologia Medica, Palermo, Sicily
  - Azienda ospedaliero-universitaria careggi, Sezione di radioterapia del dipartimento di fisiopatolo, Florence, Tuscany
  - A.O. Universitaria Pisana; Oncologia, Pisa, Tuscany
- Mexico (2):
  - Oaxaca Site Management Organization, Oaxaca City
  - Centro Oncológico Estatal; ISSSEMYM Oncología, Toluca
- Vu Medisch Centrum; Afdeling Maag-, Darm- En Leverziekte, Amsterdam, Netherlands
- Peru (4):
  - Hospital Nacional Carlos Alberto Seguin Escobedo-Essalud; Oncology & Haemathology, Arequipa
  - Hospital Nacional Edgardo Rebagliati Martins, Jesus Maria
  - Clinica Anglo Americana - Centro de Investigacion Oncologia CAA, Lima
  - Unidad de Investigacion Oncologia Clinica - Piura; Unidad de Oncología Clínica, Piura
- Poland (5):
  - Szpital Specjalistyczny Podkarpacki Ośrodek Onkologiczny, Brzozów
  - Wojewodzki Szpital Zespolony; Oddzial Chemioterapii, Elblag
  - Wojewodzkie Centrum Onkologii, Gdansk
  - COZL Oddzial Onkologii Klinicznej z pododdzialem Chemioterapii Dziennej, Lublin
  - Wojewodzki Sziptal Specjalistyczny Im. Janusza Korczaka; Oddzial Onkologiczny, Oddzial Chemioterapii, Słupsk
- Romania (8):
  - Spitalul Clinic Sf. Maria; Departmental De Oncologie, Bucharest
  - Institut of Oncology Al. Trestioreanu Bucharest; Oncology Department, Bucharest
  - Institute Of Oncology Bucharest; Medical Oncology, Bucharest
  - Cluj Clinical County Hospital; Oncology Dept, Cluj-Napoca
  - Prof. Dr. I. Chiricuta Institute of Oncology, Cluj-Napoca
  - Medisprof SRL, Cluj-Napoca
  - Municipal Clinical Hospital Filantropia; Oncology, Craiova
  - Euroclinic Center of Oncology SRL, Iași
- Russia (7):
  - Regional Oncology Hospital of Krasnodar; Oncology, Krasnodar
  - Blokhin Cancer Research Center; Combined Treatment, Moscow
  - Semashko Central Clinical Hospital; Dept of Chemotherapy, Moscow
  - GUZ Perm Region Oncology Dispensary, Perm
  - S.-Peterburg Pavlov State Medical University ; Haematology, Saint Petersburg
  - Saint-Petersburg City Clinical Oncology Dispensary, Saint Petersburg
  - SBI of Healthcare of Stavropol region Stavropol Regional Clinical Oncology Dispensary, Stavropol
- South Korea (4):
  - Severance Hospital, Seoul
  - Seoul National University Hosp; Dept Internal Med Hem Onc, Seoul
  - Asan Medical Center, Uni Ulsan Collegemedicine; Dept.Internal Medicine / Divisionhematology/Oncology, Seoul
  - Korea University Guro Hospital; Oncology, Seoul
- Spain (29):
  - Hospital Clinica Benidorm, Benidorm, Alicante
  - Complejo Hospitalario Torrecardenas; Servicio de Oncologia, Almería, Almeria
  - Consorci Hospitalari de Terrassa, Terrassa, Barcelona
  - Hospital Provincial de Castellón, Castellon, Castellon
  - Fundacion Hospital de Alcorcon; Servicio de Oncologia, Alcorcón, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Universitario de Canarias;servicio de Oncologia, San Cristóbal de La Laguna, Tenerife
  - Complejo Hospitalario Nuestra Señora de la Candelaria; Servicio de Oncologia, Santa Cruz de Tenerife, Tenerife
  - Hospital de Sagunto; Servicio de Oncologia, Sagunto, Valencia
  - Hospital de Basurto; Servicio de Oncologia, Bilbao, Vizcaya
  - Hospital Clinic i Provincial; Servicio de Farmacia, Barcelona
  - Institut Catala d Oncologia Hospital Duran i Reynals, Barcelona
  - Hospital Juan Ramon Jimenez;Servicio de Oncologia, Huelva
  - Complejo Asistencial Universitario de Leon; Servicio de Oncologia, León
  - Hospital General Universitario Gregorio Marañon; Servicio de Oncologia, Madrid
  - Hospital Ruber Internacional;Servicio de Oncologia, Madrid
  - Fundacion Jimenez Diaz; Servicio de Oncologia, Madrid
  - Hospital La Paz, Madrid
  - Complejo Hospitalario de Pontevedra; Servicio de Oncologia, Pontevedra
  - Hospital Clinico Universitario de Salamanca; Servicio de Oncologia, Salamanca
  - Hospital Universitario Virgen Macarena; Servicio de Oncologia, Seville
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Univ. Nuestra Señora de Valme;, Seville
  - Hospital Sant Pau i Santa Tecla, Tarragona
  - Complejo Hospitalario de Toledo- H. Virgen de la Salud; Servicio de Oncologia, Toledo
  - Instituto Valenciano Oncologia; Oncologia Medica, Valencia
  - Hospital Clinico Universitario de Valencia; Servicio de Onco-hematologia, Valencia
  - Hospital Universitario la Fe; Servicio de Oncologia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Thailand (5):
  - Phramongkutklao Hospital;Dept Surgery/Surgical Oncology Unit, Bangkok
  - Ramathibodi Hospital; Department of Surgery/Breast and Endocrine Unit, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital; Department of Surgery/Head Neck and Breast Unit; Clinical Trial, Chiang Mai
  - Srinagarind Hospital; Department of Surgery, Khon Kaen
  - Songklanagarind Hospital; Department of Surgery, Songkhla
- United Kingdom (10):
  - Royal Bournemouth General Hospital; Oncology, Bournemouth
  - Velindre Cancer Centre; Oncology Dept, Cardiff
  - Broomfield Hospital, Chelmsford
  - University Hospital of North Durham; Oncology, Durham
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Christie Hospital; Breast Cancer Research Office, Manchester
  - Nottingham City Hospital, Nottingham
  - Peterborough City Hospital, Edith Cavell Campus; Oncology Department, Peterborough
  - Great Western Hospital; Clinical Oncology, Swindon
  - Royal Cornwall Hospital; Dept of Clinical Oncology, Truro

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 452 participants were randomized to one of two treatment arms: trastuzumab and capecitabine (Arm A, 224 participants) or pertuzumab with trastuzumab and capecitabine (Arm B, 228 participants). Of participants randomized to Arm A: trastuzumab and capecitabine, 6 participants did not receive study treatment.
Groups:
- A: Capecitabine + Trastuzumab: Capecitabine [Xeloda]: 1250 mg/m2 po twice daily for 14 days every 3 weeks. Trastuzumab [Herceptin]: 8 mg/kg iv loading, then 6 mg/kg iv every 3 weeks.
- B: Capecitabine + Trastuzumab + Pertuzumab: Capecitabine [Xeloda]: 1000 mg/m2 po twice daily for 14 days every 3 weeks. Pertuzumab [Perjeta]: 840 mg iv loading, then 420 mg iv every 3 weeks. Trastuzumab [Herceptin]: 8 mg/kg iv loading, then 6 mg/kg iv every 3 weeks.
Period: Overall Study
Arm/Group | A: Capecitabine + Trastuzumab | B: Capecitabine + Trastuzumab + Pertuzumab
Started | 224 | 228
Completed | 52 | 65
Not Completed | 172 | 163
Not completed — Death | 136 | 134
Not completed — Withdrew consent or lost to follow-up | 36 | 29

BASELINE CHARACTERISTICS:
Population: This is the safety population, which includes all participants who received any amount of study drug; 6 participants randomized to the Capecitabine + Trastuzumab arm withdrew before receiving any study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | A: Capecitabine + Trastuzumab | B: Capecitabine + Trastuzumab + Pertuzumab | Total
Number analyzed (Participants) | 218 | 228 | 446
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (10.10) | 53.0 (11.21) | 54.0 (10.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 218 | 228 | 446
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Russian Federation | 8 | 3 | 11
  Argentina | 3 | 4 | 7
  Romania | 6 | 8 | 14
  Hungary | 13 | 29 | 42
  Hong Kong | 5 | 11 | 16
  United Kingdom | 18 | 17 | 35
  Thailand | 0 | 5 | 5
  Spain | 39 | 31 | 70
  Canada | 3 | 6 | 9
  Czech Republic | 12 | 10 | 22
  Austria | 2 | 3 | 5
  Netherlands | 0 | 2 | 2
  Belgium | 12 | 11 | 23
  Poland | 6 | 6 | 12
  Brazil | 7 | 6 | 13
  Korea, Republic of | 14 | 24 | 38
  Italy | 16 | 18 | 34
  Mexico | 1 | 0 | 1
  France | 19 | 12 | 31
  Peru | 7 | 8 | 15
  Germany | 23 | 11 | 34
  Croatia | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (Independent Assessment)
Description: Progression Free Survival (PFS) was defined as the time from randomization to first documented disease progression (PD), as determined by an Independent Review Facility (IRF) using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.0, or death from any cause, whichever occurred first. PD was defined as at least a 20% increase in the sum of the longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; or the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. IRF review of tumor assessment ceased after the primary PFS analysis. The primary endpoint was analyzed after approximately 337 IRF-assessed PFS events were observed.
Time Frame: Tumor assessments every 9 weeks from randomization until Week 27, then every 12 weeks thereafter, until IRF-determined PD, initiation of alternative anticancer medication, or death (up to 5.5 years).
Population: All randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A: Capecitabine + Trastuzumab | B: Capecitabine + Trastuzumab + Pertuzumab
Number analyzed (Participants) | 224 | 228
months | 9.0 [8 to 10] | 11.1 [9 to 13]
Statistical Analysis 1: Comparison: A: Capecitabine + Trastuzumab vs B: Capecitabine + Trastuzumab + Pertuzumab; The null hypothesis for the primary endpoint is that the survival distributions of IRF-assessed PFS in the two treatment groups are the same. The alternative hypothesis is that the survival distributions of IRF-assessed PFS in the treatment and the control arms are different: H0: IRF PFS<pertuzumab> = IRF PFS<control> vs. H1: IRF PFS<pertuzumab> ≠ IRF PFS<control>; Test type: Superiority; p = 0.0731, Log Rank — The primary endpoint, IRF-assessed PFS, is tested at a two-sided 5% significance level; Two-sided and stratified by: prior CNS disease present/absent, measurable disease at baseline, and response to trastuzumab in 1L metastatic setting; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.65 to 1.02] — The stratified Cox proportional hazard model will be used to estimate the HR between the two treatment arms and its 95% CI

2. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) was defined as the time from the date of randomization to the date of death from any cause. The results of the final OS analysis are presented here. Participants who were alive or lost to follow-up at the time of the analysis were censored at the last known alive date. Participants with no postbaseline information were censored at the time of randomization plus 1 day. Prior to the final data analysis cut-off, it was ensured that all participants who were in survival follow-up had been contacted as recently as possible within the last 3 months to confirm current survival status.
Time Frame: From randomization until death from any cause (up to 7.5 years).
Population: All randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | A: Capecitabine + Trastuzumab | B: Capecitabine + Trastuzumab + Pertuzumab
Number analyzed (Participants) | 224 | 228
Months | 28.1 [22 to 35] | 37.2 [33 to 42]

3. Secondary Outcome: Overall Survival (OS) Rate Based on a 2-year Truncated Analysis
Description: The Overall Survival (OS) 2-year truncated analysis is the Kaplan-Meier estimate of the percentage of participants who were surviving at 2 years. OS is defined as the time from the date of randomization to the date of death from any cause, with censoring of all events and follow-up beyond the end of the second year.
Time Frame: From randomization until death from any cause (up to 2 years)
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Capecitabine + Trastuzumab | B: Capecitabine + Trastuzumab + Pertuzumab
Number analyzed (Participants) | 224 | 228
Percentage of participants | 55.0 [48.07 to 61.85] | 74.9 [69.05 to 80.68]

4. Secondary Outcome: Investigator Assessment Progression-Free Survival (PFS)
Description: Investigator Assessment Progression-Free Survival (PFS) was defined as the time from randomization to the first documented progressive disease, as determined by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST) v1.0, or death from any cause, whichever occurred first. PD is defined as at least a 20% increase in the sum of the longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; or the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Tumor assessments every 9 weeks from randomization until Week 27, then every 12 weeks thereafter, until IRF-determined PD, initiation of alternative anticancer medication, or death (up to 7.5 years).
Population: All randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | A: Capecitabine + Trastuzumab | B: Capecitabine + Trastuzumab + Pertuzumab
Number analyzed (Participants) | 224 | 228
Months | 9.0 [8 to 12] | 11.8 [9 to 14]

5. Secondary Outcome: Time to Progression (TTP) Based Upon Independent Review Facility (IRF) Assessment
Description: Time to Progression (TTP) was defined as time between randomization and the first occurrence of progressive disease (PD), based on IRF assessment.
Time Frame: as for outcome 1
Population: All randomized participants.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | A: Capecitabine + Trastuzumab | B: Capecitabine + Trastuzumab + Pertuzumab
Number analyzed (Participants) | 224 | 228
Weeks | 39.0 [35 to 44] | 50.6 [39 to 62]

6. Secondary Outcome: Time to Treatment Failure (TTF) Based Upon Independent Review Facility (IRF) Assessment
Description: Time to Treatment Failure (TTF) was defined as time between randomization and date of disease progression based on independent review, death, or withdrawal of treatment due to adverse events, withdrawn informed consent, refusal of treatment/failure to cooperate, or failure to return, whichever occurred first.
Time Frame: as for outcome 1
Population: All randomized participants.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | A: Capecitabine + Trastuzumab | B: Capecitabine + Trastuzumab + Pertuzumab
Number analyzed (Participants) | 224 | 228
Weeks | 39.0 [34 to 44] | 50.9 [39 to 62]

7. Secondary Outcome: Overall Objective Response Rate (ORR)
Description: Overall Objective Response Rate is based upon investigator and IRF assessments. Objective Response Rate (ORR) was defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR) among those who had measurable disease at baseline. CR was defined as the disappearance of all target lesions. PR was defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
Time Frame: as for outcome 1
Population: Participants without a post-baseline tumor assessment were considered to be non-responders and were not included in this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | A: Capecitabine + Trastuzumab | B: Capecitabine + Trastuzumab + Pertuzumab
Number analyzed (Participants) | 164 | 163
Percentage of participants
  Complete Response (CR) - IRF Assessment | 0 | 1.8
  Partial Response (PR) - IRF assessment | 32.9 | 38.7
  Complete Response (CR) - Investigator Assessed | 1.2 | 6.7
  Partial Response (PR) - Investigator Assessed | 36.0 | 38.0

8. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Clinical Benefit Rate is based upon Independent Review Facility (IRF) assessments; defined as the percentage of participants a complete response (CR), partial response (PR), or stable disease for at least 8 cycles or 6 months.
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Capecitabine + Trastuzumab | B: Capecitabine + Trastuzumab + Pertuzumab
Number analyzed (Participants) | 224 | 228
Percentage of participants | 54.0 [47.3 to 60.7] | 63.6 [57.0 to 69.8]

9. Secondary Outcome: Duration of Objective Response
Description: Duration of Objective Response was defined for the subpopulation of responders as time from first Independent Review Facility (IRF)-assessed complete response (CR) or partial response (PR) to subsequent first documented, IRF-confirmed evidence of disease progression. Only participants with an objective response were included in the analysis of duration of objective response.
Time Frame: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | A: Capecitabine + Trastuzumab | B: Capecitabine + Trastuzumab + Pertuzumab
Number analyzed (Participants) | 54 | 66
Weeks | 30.0 [21 to 42] | 51.6 [42 to 57]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded and reported during the study and up to two years after the last dose of the study drug was received.
Arm/Group | A: Capecitabine + Trastuzumab | B: Capecitabine + Trastuzumab + Pertuzumab
All-Cause Mortality (participants affected / at risk) | 136/218 | 134/228
Serious Adverse Events (participants affected / at risk) | 53/218 | 58/228
Other Adverse Events (participants affected / at risk) | 209/218 | 216/228
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: Capecitabine + Trastuzumab (N=218) | B: Capecitabine + Trastuzumab + Pertuzumab (N=228)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 8 (8)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Left Ventricular Dysfunction (Cardiac disorders) | 4 (4) | 13 (13)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Angina Unstable (Cardiac disorders) | 0 (0) | 1 (1)
Arteriospasm Coronary (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Femur Fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Acetabulum Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bone Fissure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Craniocerebral Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint Dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meniscus Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Synovial Rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Catheter Site Infection (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium Difficile Colitis (Infections and infestations) | 0 (0) | 1 (1)
Device Related Infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Phlebitis Infective (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pulmonary Tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Secondary Cerebellar Degeneration (Nervous system disorders) | 1 (1) | 0 (0)
Status Epilepticus (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (4)
Pulmonary Thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
General Physical Health Deterioration (General disorders) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 2 (2) | 2 (2)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Device Related Thrombosis (General disorders) | 0 (0) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vena Cava Thrombosis (Vascular disorders) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis Superficial (Vascular disorders) | 1 (1) | 0 (0)
Venous Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acute Promyelocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cervix Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Retinal Detachment (Eye disorders) | 0 (0) | 1 (1)
Anaphylactic Shock (Immune system disorders) | 0 (0) | 1 (1)
Blood Sodium Decreased (Investigations) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Ureteric Stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Endometrial Hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: Capecitabine + Trastuzumab (N=218) | B: Capecitabine + Trastuzumab + Pertuzumab (N=228)
Diarrhoea (Gastrointestinal disorders) | 128 (275) | 157 (436)
Nausea (Gastrointestinal disorders) | 97 (152) | 88 (129)
Vomiting (Gastrointestinal disorders) | 45 (56) | 37 (58)
Stomatitis (Gastrointestinal disorders) | 32 (39) | 41 (60)
Abdominal Pain (Gastrointestinal disorders) | 30 (36) | 28 (50)
Abdominal Pain Upper (Gastrointestinal disorders) | 24 (31) | 29 (45)
Dyspepsia (Gastrointestinal disorders) | 22 (23) | 24 (33)
Constipation (Gastrointestinal disorders) | 21 (27) | 18 (22)
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 159 (242) | 129 (179)
Rash (Skin and subcutaneous tissue disorders) | 11 (12) | 35 (45)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (7) | 21 (29)
Dry Skin (Skin and subcutaneous tissue disorders) | 9 (10) | 16 (17)
Nail Disorder (Skin and subcutaneous tissue disorders) | 8 (8) | 14 (15)
Alopecia (Skin and subcutaneous tissue disorders) | 11 (12) | 6 (6)
Asthenia (General disorders) | 51 (87) | 47 (77)
Fatigue (General disorders) | 39 (59) | 44 (62)
Mucosal Inflammation (General disorders) | 27 (36) | 32 (45)
Pyrexia (General disorders) | 20 (24) | 29 (41)
Oedema Peripheral (General disorders) | 13 (13) | 18 (19)
Chest Pain (General disorders) | 12 (15) | 9 (11)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 15 (24) | 27 (32)
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 (19) | 21 (27)
Back Pain (Musculoskeletal and connective tissue disorders) | 18 (23) | 20 (23)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 12 (20) | 17 (21)
Bone Pain (Musculoskeletal and connective tissue disorders) | 12 (16) | 8 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (8) | 12 (19)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 5 (7) | 12 (13)
Headache (Nervous system disorders) | 39 (68) | 40 (52)
Dizziness (Nervous system disorders) | 21 (28) | 24 (26)
Neuropathy Peripheral (Nervous system disorders) | 14 (17) | 16 (17)
Paraesthesia (Nervous system disorders) | 13 (15) | 9 (9)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 12 (15) | 25 (37)
Urinary Tract Infection (Infections and infestations) | 17 (20) | 21 (28)
Upper Respiratory Tract Infection (Infections and infestations) | 9 (12) | 19 (46)
Paronychia (Infections and infestations) | 11 (15) | 15 (16)
Influenza (Infections and infestations) | 4 (5) | 12 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 22 (27) | 30 (38)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 24 (28) | 21 (25)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 12 (14)
Decreased Appetite (Metabolism and nutrition disorders) | 28 (43) | 36 (43)
Hypokalaemia (Metabolism and nutrition disorders) | 13 (19) | 28 (40)
Neutropenia (Blood and lymphatic system disorders) | 38 (89) | 29 (74)
Anaemia (Blood and lymphatic system disorders) | 17 (23) | 21 (28)
Weight Decreased (Investigations) | 13 (14) | 19 (20)
Aspartate Aminotransferase Increased (Investigations) | 11 (15) | 17 (26)
Alanine Aminotransferase Increased (Investigations) | 8 (11) | 17 (24)
Insomnia (Psychiatric disorders) | 12 (17) | 23 (27)
Hypertension (Vascular disorders) | 14 (18) | 19 (19)
Lacrimation Increased (Eye disorders) | 13 (17) | 6 (8)
Left Ventricular Dysfunction (Cardiac disorders) | 5 (5) | 13 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.